CLINICAL TRIAL: NCT03550768
Title: Effect of Anatomy of Major Duodenal Papilla on the Difficulty of Cannulation During Endoscopic Retrograde Cholangiopancreatography (ERCP)
Brief Title: Effect of Anatomy of Major Duodenal Papilla on the Difficulty of Cannulation During Endoscopic Retrograde Cholangiopancreatography
Status: Completed | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Collaborators: The Second Affiliated Hospital of Chongqing Medical University (Other); Huaihe Hospital of Henan University (Other); Successful Hospital of Xiamen university (Unknown)
Responsible Party: Principal Investigator, Yanglin Pan, Associate Professor, Air Force Military Medical University, China
Other Study IDs: KY20180081-2
Record Dates: First submitted 2018-05-16; First posted 2018-06-08 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Pancreaticobiilary Diseases; Endoscopic Retrograde Cholangiopancreatography
Keywords: ERCP; anatomy of major duodenal papilla

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MDP: ERCP was performed by trainees or trainers. Before the cannulation, the photo of major duodenal papilla will be taken carefully to evaluate its size, morphology, orientation and location. All patients initially received wire-guided cannulation with a sphincterotome, If cannulation failed, precut sphincterotomy or the double-wire technique was performed when appropriate. Therapeutic manipulation (eg, sphincterotomy, balloon dilation, stone extraction, and stenting) was done when appropriate. Pancreatic duct stent placement was performed at the discretion of the endoscopists.
  Interventions: Other: MDP

INTERVENTIONS:
Other: MDP — evaluate the anatomy of each major duodenal papilla before selective cannulation during ERCP

SUMMARY:
Selective cannulation is an essential step for the success of ERCP. The successful cannulation is influenced by types of disease (such as Sphincter of Oddi Dysfunction and duodenal stricture), the experience of endoscopists and the anatomy of papilla. It is suggested that the size, morphology, orientation and location of major duodenal papilla (MDP), could cause a difficult cannulation (Endoscopy 2016; 48: 657-683). However, the related evidences are limited. The investigators hypothesized that special anatomy of papilla, such as a lanky shape (defined by the higher ratio of length to width) and a deeper location, could increase the difficulty of cannulation. Here the investigators investigated the effects of the anatomy of major duodenal papilla on post-ERCP pancreatitis and the procedure of cannulation in patients undergoing ERCP.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80
* Patients with native papilla who underwent ERCP

Exclusion Criteria:

* Prior endoscopic sphincterotomy
* Minor pancreatic duct as the targeted duct
* History of prior upper gastrointestinal surgery, such as Billroth I, II and Roux-en-Y
* Fistula of MDP
* Papillary carcinoma or adenoma
* Duodenal obstruction, type II
* Prior stent placement in common bile duct or pancreatic duct
* Pregnant or breastfeeding women
* Unwilling or inability to provide consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with native papilla who underwent ERCP
Sampling Method: Probability Sample
Enrollment: 658 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
post-ERCP pancreatitis incidence | 48 hours
  frequency of post-ERCP pancreatitis

SECONDARY OUTCOMES:
Rate of difficult cannulation | 3 hours
  difficult cannulation was defined as when total cannulation time was more than 5minutes, total cannulation attempts more than 5 times or inadvertent pancreatic duct cannulation more than 1 time.
Cannulation attempts | 3 hours
  the sphincterotome touching the papilla for at least 5 seconds will be considered as one attempt.
Total cannulation time | 3 hours
  the time from the moment the sphincterotome touch the papilla to the guide wire advance into the target duct.
Unintended pancreatic duct cannulation | 3 hours
  the guide wire unintentionally entered into the undesired pancreatic duct
Complication rate | 48 hours
  frequency of any adverse outcome that required hospital admission or prolonged hospital stay necessary for management of the complication, including pancreatitis, bleeding, biliary infection or perforation.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Department of gastroenterology, Successful Hospital of Xiamen university, Xiamen, Fujian
  - Huaihe Hospital of Henan University, Kaifeng, Henan
  - Endoscopic center, Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi
  - Department of gastroenterology, Second Affiliated Hospital of Chongqing Medical University, Chongqing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang X, Zhao J, Wang L, Ning B, Zeng W, Tao Q, Ren G, Liang S, Luo H, Wang B, Farrell JJ, Pan Y, Guo X, Wu K. Relationship between papilla-related variables and post endoscopic retrograde cholangiopancreatography pancreatitis: A multicenter, prospective study. J Gastroenterol Hepatol. 2020 Dec;35(12):2184-2191. doi: 10.1111/jgh.15135. Epub 2020 Jun 29. PMID 32511794